CLINICAL TRIAL: NCT02786303
Title: Interest of Whole-body MRI Correlated to Spreading Sequences for Staging
Brief Title: Interest of Whole-body MRI Correlated to Spreading Sequences for Staging Neuroendocrine Tumors
Acronym: LAB-2013-01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI13103
Record Dates: First submitted 2016-05-12; First posted 2016-06-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Neuroendocrine Tumors With Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- arm whole-body MRI (Other)
  Interventions: Device: Whole-body diffusion- weighted MRI

INTERVENTIONS:
Device: Whole-body diffusion- weighted MRI

SUMMARY:
The diagnosis and the follow-up of neuroendocrine tumors can be difficult to assess, especially in the detection of metastasis as they can grow in different organs such as liver, lungs, bones or lymph nodes. Nowadays, the diagnosis is made with two main imaging techniques which are the thoraco-abdomino-pelvic CT-scan and a scintigraphic method (Octreoscan and sometimes a TEP-scan). The use of a whole-body MRI is more and more often used for the detection and evaluation of tumors and metastases; therefore, it could be used for neuroendocrine tumors. The MRI would allow to replace the two imaging techniques and to avoid the use of irradiation but also to have a better detection of metastases. This purpose of the study was to evaluate this statement by assessing the consistency between the routine techniques and the MRI and finally to update the recommendation if the study is positive.

DETAILED DESCRIPTION:
The main metastatic sites of neuroendocrine tumors can be the liver, the bones, the lungs and lymph nodes. According to the French recommendations (" Thesaurus national de cancérologie digestive "), the initial assessment includes a thoraco-abdomino-pelvic CT-scan and a scintigraphic method (Octreoscan and TEP-scan if Octreoscan negative). The aim is to detect metastases and tumoral progression to offer the appropriate treatment, such as surgery. Due to its high contrast resolution, its absence of irradiation, and diffusion sequences, the MRI is more and more used to detect tumor progression. The recent literature shows better results with the diffusion sequences than the T2-weighted sequences and, potentially, than the contrast-enhanced sequences to detect liver metastasis. The whole-body diffusion-weighted MRI seems promising for the staging and the following of some cancers. Only two publications have evaluated the diagnostic value of diffusion sequences to detect pancreatic neuroendocrine tumors and liver metastasis. Yet, no publication has assessed the diagnostic value of whole-body diffusion-weighted MRI in the patients with neuroendocrine tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderately to well-differentiated neuroendocrine tumors with stage ≥ 3 according to the classification ENETS, regardless the tumor site and the OMS
* Patients who signed the informed consent
* Patients followed in one of the participating center

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Correspondance between whole-body diffusion-weighted MRI and thoraco-abdomino-pelvic CT-scan associated with a scintigraphic method in the detection and staging of neuroendocrine tumors and metastases | Day 1

REFERENCES:
- [Derived] Minon M, Soriano C, Morland D, Walter T, Lepage C, Tabarin A, Deblock M, Rousset P, Barbe C, Hoeffel C, Cadiot G. Prospective comparison of whole-body MRI with diffusion-weighted and conventional imaging for the follow-up of neuroendocrine tumors. Endocrine. 2020 Jan;67(1):243-251. doi: 10.1007/s12020-019-02095-5. Epub 2019 Sep 28. PMID 31564038